CLINICAL TRIAL: NCT00447161
Title: Bacillus Clausii in Preventing Antibiotic-Associated Diarrhea Among Filipino Infant and Children: A Multi-Center, Randomized, Open-Label Controlled (Treatment vs No Treatment) Clinical Trial of Efficacy and Safety
Brief Title: Preventing Antibiotic-Associated DiarRhea Using Erceflora
Acronym: PADRE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Medical Affairs Study Director, sanofi-aventis
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ENTER_L_01125
Record Dates: First submitted 2007-03-13; First posted 2007-03-14 (Estimated); Last update posted 2008-09-05 (Estimated); Status verified 2008-09

CONDITIONS: Diarrhea, Infantile
MeSH Terms: conditions — Diarrhea, Infantile

ARMS (2):
- 1 (Experimental): Bacillus Clausii Multi ATB Resist
  Interventions: Drug: Bacillus Clausii Multi ATB Resist
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Bacillus Clausii Multi ATB Resist — Twice daily dose of 1 vial of 1x10^9 of Bacillus clausii spores, orally suspension in water
  Arms: 1
Drug: Placebo — Matched placebo
  Arms: 2

SUMMARY:
To determine the effectiveness of the pre-biotic Bacillus clausii in preventing antibiotic associated diarrhea among hospitalized immunocompetent Filipino children.

ELIGIBILITY:
Inclusion Criteria:

* Clinically stable children with mild to moderate illness admitted for treatment of bacterial infection.

Exclusion Criteria:

* Children with unstable medical condition
* In any form of immunocompromized state
* With contraindication to take medication
* Has taken antibiotics for 3 weeks before start of trial.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 6 Months to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 323 (Actual)
Dates: Start 2006-07; Primary Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Reduction in the incidence of antibiotic-associated diarrhea (relative risk) | From baseline to end of treatment
All adverse event regardless of seriousness or relationship to the study drug | From baseline to end of treatment

SECONDARY OUTCOMES:
Reduction in the number of antibiotic-associated diarrhea events per day | From baseline to end of treatment
Reduction in the severity of diarrhea events | From baseline to end of treatment
Reduction in Gastrointestinal-related symptoms (nausea, vomiting, abdominal pain)over-all reduction in the number of hospitalization days beween control and treatment groups. | From baseline to end of treatment
Reduction in C. dificille -associated diarrhea. | From baseline to end of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Paz Figueroa, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis, Manila, Philippines